CLINICAL TRIAL: NCT02504073
Title: Clinical Reasoning Process of Physiotherapists When Observing Hemiplegic Gait
Status: Completed | Type: Observational
Sponsor: Technical University of Bern (Other)
Responsible Party: Principal Investigator, Clare Maguire, MPTSc (cand) PhD, Technical University of Bern
Other Study IDs: EKNZ08/12/14
Record Dates: First submitted 2015-07-15; First posted 2015-07-21 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Stroke
Keywords: Clinical Reasoning; Physiotherapists
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PT's working in stroke in NW-Switzerland: 54 Physiotherapists (PT's) working in north-west Switzerland (at Bruderholzspital, RehaB Basel, Klinik Tschugg, Reha Rheinfelden, RehaClinic Zurzach) are asked to analyse videos of 6 hemiplegic patients when walking. They are asked to write down their main observations, the major problem and hypotheses about how this major problem is produced.
  There is no intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The goal of this study is to find out what clinical reasoning process physiotherapists undergo when observing hemiplegic patients gait.

DETAILED DESCRIPTION:
Physiotherapists don't usually use any assessments to evaluate gait but observe it without an instrument. The questions in this study are:

* what abnormalities can physiotherapists detect when observing a patient walking?
* what do they consider the main problem that has a negative effect on the patient's walking?
* what hypothesis do they generate?
* how is the inter-rater reliability for the "main problem" and the hypothesis?

ELIGIBILITY:
Inclusion criteria:

* chartered physiotherapists
* physiotherapists in training
* working with stroke patients

Exclusion criteria:

- other languages than German

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: physiotherapists working with stroke patients
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-03; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Groups:
- PT's Working With Stroke Patients in NW-Switzerland: Physiotherapists from Bruderholzspital, RehaB Basel, Klinik Tschugg, Reha Rheinfelden, RehaClinic Zurzach
Period: Overall Study
Arm/Group | PT's Working With Stroke Patients in NW-Switzerland
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | PT's Working With Stroke Patients in NW-Switzerland
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 54
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Gait Abnormalities Observed
Description: The questionnaire will be the basis of this study as it will be the basis for open coding. It is handed out to 54 observers (=physiotherapists) and will be filled in 6 times (for 6 patient videos).
  The questionnaire consists of 3 main questions:
  1. what gait abnormalities do you see?
  2. What do you consider the main problem (1 sentence)
  3. what is your hypothesis (max. 3) The question one delivers different items (each new observation is a new item) that were determined patient by patient and rater by rater by three independent researchers. They were then listed and categorised by consensus. Finally, the frequency of each item was analysed globally and for each patient.
Time Frame: up to 2 months
Measure: Number; unit: number of different gait abnormalities
Arm/Group | PT's Working With Stroke Patients in NW-Switzerland
Number analyzed (Participants) | 54
number of different gait abnormalities | 177

2. Primary Outcome: Number of Main Problems Observed
Description: This outcome is a result of the second part of the Questionnaire: 1) What Gait Abnormalities do You See? 2) What do You Consider the Main Problem (1 Sentence) 3) What is Your Hypothesis (Max. 3) By consensus the three independent researchers identified the main statements from the sentences written. Items were afterwards categorised. Finally the frequency of each item was analysed globally and for each patient.
Time Frame: up to 2 months
Measure: Number; unit: number of different main problems
Groups:
- PT's Working in Stroke in NW-Switzerland: 54 Physiotherapists from Bruderholzspital, RehaB Basel, Klinik Tschugg, Reha Rheinfelden, RehaClinic Zurzach are asked to analyse videos of 6 hemiplegic patients when walking. They are asked to write down their main observations, the major problem and hypotheses about how this major problem is produced.
  There is no intervention.
  No intervention: No intervention
Arm/Group | PT's Working in Stroke in NW-Switzerland
Number analyzed (Participants) | 54
number of different main problems | 93

3. Primary Outcome: Number of Hypotheses Observed
Description: This outcome is a result of the third part of the questionnaire: 1) What Gait Abnormalities do You See? 2) What do You Consider the Main Problem (1 Sentence) 3) What is Your Hypothesis (Max. 3) By consensus the three independent researchers identified and categorised all the listed hypotheses from question number three of the questionnaire. After that the use frequency of each item was analysed globally and for each patient.
Time Frame: up to 2 months
Measure: Number; unit: Number of different hypotheses
Arm/Group | PT's Working in Stroke in NW-Switzerland
Number analyzed (Participants) | 54
Number of different hypotheses | 119

ADVERSE EVENTS:
Time Frame: 1 year
Description: No adverse events are to be expected as intervention group were physiotherapists that, over the period of 2 hours, analysed 6 videos of patients walking.
Arm/Group | PT's Working With Stroke Patients in NW-Switzerland
All-Cause Mortality (participants affected / at risk) | 0/54
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 0/54

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes